CLINICAL TRIAL: NCT01809171
Title: Placebo-controlled Trial With Vitamin D to Prevent Worsening/Relieve Aromatase Inhibitor-induced Musculoskeletal Symptoms in Breast Cancer Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inclusion problems
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: s55283; 2013-001064-27 (EudraCT Number)
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Musculoskeletal Disease
MeSH Terms: conditions — Breast Neoplasms; Musculoskeletal Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D3 (Experimental): 1000 mg Ca2+/800IU vitamin D3 daily + 25 000IU vitamin D3 weekly during 6 months
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): 1000 mg Ca2+/ 800IU vitamin D3 daily + 25000IU placebo every week during 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — ampoule
  Arms: vitamin D3
Drug: Placebo — ampoule
  Arms: Placebo

SUMMARY:
The third generation oral aromatase inhibitors (AIs) are increasingly being used in the management of estrogen receptor positive breast cancer. One of the issues related with administration of oral AIs is their side effects, particularly on the musculoskeletal system. Although the prevalence and importance of arthralgia and myalgia occurring in BC patients receiving adjuvant AIs are evident, the mechanisms clearly explaining these invalidating symptoms are unknown.

In this project, we aim to unravel the interaction between vitamin D and musculoskeletal adverse events experienced by AI users. We will also evaluate how vitamin D supplementation affects AI-induced musculoskeletal symptoms in breast cancer patients, by means of a randomized placebo-controlled double blind clinical trial. We will assess changes in the musculoskeletal system by using magnetic resonance imaging of joints, hand grip strength and also monitor serum IGF-I and estrogen levels together with bone resorption and formation markers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status
* Currently being treated with an AI in the adjuvant setting (minimum for 8 weeks)
* AIMSS as determined by new or worsened musculoskeletal complaints following AI therapy
* Vitamin D deficiency (<30ng/ml)
* Caucasian

Exclusion Criteria:

* Hormone replacement therapy last 6 months
* Current use or in the last 12 months of bisphosphonates
* Tamoxifen use in last 6 months
* History of kidney stones
* History of hypercalcemia/hypercalciuria or hyperthyroidism
* Paget's disease of the bone
* Current use of Digitalis/digoxin or thiazide diuretics
* Current use of vitamin D (or multivitamin) supplementation should be stopped

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in musculoskeletal pain and 250HD levels | 3 monthly during one year

SECONDARY OUTCOMES:
Change from baseline in bone parameters, estrogen and IGF-I levels and fluid accumulation and tendon pathologies, as seen on MRI | 3 monthly during 1 year, MRI at baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Roberts KE, Adsett IT, Rickett K, Conroy SM, Chatfield MD, Woodward NE. Systemic therapies for preventing or treating aromatase inhibitor-induced musculoskeletal symptoms in early breast cancer. Cochrane Database Syst Rev. 2022 Jan 10;1(1):CD013167. doi: 10.1002/14651858.CD013167.pub2. PMID 35005781